CLINICAL TRIAL: NCT06329180
Title: Evaluation of the Knowledge, Attitudes and Behaviours of Health Professionals Regarding Physical Activity and Metabolic Health Screening for People With Mental Illness
Brief Title: Exercise in Mental Illness Questionnaire: French Validation
Status: Enrolling by invitation | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Davy Vancampfort, Professor, KU Leuven
Other Study IDs: 26.02.2024
Record Dates: First submitted 2024-03-19; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The validation of the French version of the Exercise in Mental Illness Questionnaire - Health Practitioner Version (EMIQ-HP) is a prospective observational case-only study involving: (a) translation to French, (b) an expert consensus meeting with French speaking experts from Canada to reach a first version, (c) back translation to English, (d) evaluation of the back-translation by the original authors of the EMIQ-HP, (e) an expert consensus meeting with French speaking experts from Canada to reach a final version based on comments of the original authors, and (f) test-retest reliability study. Test-retest reliability will be analysed through two points of measurement with an interval of 7 days.

DETAILED DESCRIPTION:
The aim of this study is to cross-culturally validate the French translation of the Exercise in Mental Illness Questionnaire - Health Practitioner version (EMIQ-HP) scale and investigate the test-retest reliability. We hypothesize that the French validated translation of the Exercise in Mental Illness Questionnaire - Health Practitioner version (EMIQ-HP) scale will show and excellent test - retest reliability. National and international experts from Belgium, Canada and Switzerland are requested to join the expert panel and requested to be available on 2 different occasions, i.e. following the first translation and following the feedback of the original authors on the back translation in order to reach consensus on the final version. For the test-retest part of this study, all health care providers of the Centre Hospitalier Psychiatrique Chêne aux Haies (i.e. nurses, psychologists, physiotherapists, somatic medical doctors, psychiatrists) will be invited to participate. Following written informed consent procedure, participants will complete the EMIQ-HP which will be completed a second time exactly one week following the first completion

ELIGIBILITY:
National and international experts from Belgium and Canada will be requested to join the expert panel and requested to be available on 2 different occasions, i.e. following the first translation and following the feedback of the original authors on the back translation in order to reach consensus on the final version. For the test-retest part of this study, all health care providers of the Centre Hospitalier Psychiatrique Chêne aux Haies (i.e. nurses, psychologists, physiotherapists, somatic medical doctors, psychiatrists) will be invited to participate. There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: National and international experts from Belgium and Canada will be requested to join the expert panel and requested to be available on 2 different occasions, i.e. following the first translation and following the feedback of the original authors on the back translation in order to reach consensus on the final version. For the test-retest part of this study, all health care providers of the Centre Hospitalier Psychiatrique Chêne aux Haies (i.e. nurses, psychologists, physiotherapists, somatic medical doctors, psychiatrists) will be invited to participate. There are no specific exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Intra-class-correlation coefficients (ICC 3,1 | 7 days test -retest
  EMIQ items

CONTACTS AND LOCATIONS:
Overall Officials: Davy Vancampfort, Phd, Principal Investigator — KU Leuven
Locations (1):
- Centre Hospitalier Psychiatrique Chêne aux Haies, Mons, Belgium

IPD SHARING:
Plan to Share IPD: No